CLINICAL TRIAL: NCT04291846
Title: A Randomized, Open, Single-center, Two-cycle, Double-sequence Crossover Study to Investigate the Effects of a High-fat Diet on the Pharmacokinetics of Healthy Chinese Adult Subjects After Oral Administration of SHR1459 Tablets
Brief Title: A Food Effect Study of SHR1459 on Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SHR1459-I-103
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-05

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Diet, High-Fat; P-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: SHR1459 fasted in P1, high-fat diet in P2
- B (Experimental)
  Interventions: Drug: SHR1459 high-fat diet in P1, fasted in P2

INTERVENTIONS:
Drug: SHR1459 fasted in P1, high-fat diet in P2 — SHR1459 administration in fasted condition in period 1, SHR1459 administration after high-fat diet in period 2
  Arms: A
Drug: SHR1459 high-fat diet in P1, fasted in P2 — SHR1459 administration after high-fat diet in period 1, SHR1459 administration in fasted condition in period 2
  Arms: B

SUMMARY:
The primary objective of the study is to evaluate the effect of high-fat diet on pharmacokinetics of healthy Chinese adult subjects after oral administration of SHR1459 tablets.

The secondary objective of the study is to evaluate the safety of single dose of SHR1459 orally in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18 or above (including 18 years old) at the date of signing the informed consent;
2. Male body weight ≥ 50kg, female body weight ≥ 45kg, body mass index (BMI) within the range of 19 ~ 28kg /m2 (including 19 and 28) (BMI= weight (kg)/height 2 (m2));
3. During screening period physical examination, vital signs, blood routine, urine routine, blood biochemistry, coagulation, abdominal ultrasound, chest X-ray and other examination results must be within the normal range consistent with age and gender, or in accordance with the protocol, or judged to be "no clinical significance (NCS)" if beyond the normal range;
4. The 12-lead ECG should be normal, with male QTcF < 430ms and female QTcF < 450ms; QTc interval is corrected by Fridericia formula (QTcF = QT/(RR^0.33), RR is the standardized heart rate value, calculated by dividing heart rate by 60);
5. Negative pregnancy test for women of child-bearing age;
6. Agree to abstain from sex or use effective non-drug contraceptives from screening to at least 3 months after the last study drug administration (female subjects are also required to abstain or use effective non-drug contraceptives two weeks prior to study entry);
7. The subject can communicate well with the researcher, understand and comply with the requirements of the study, understand and sign the informed consent.

Exclusion Criteria:

1. Allergic constitution or known allergy to the research drug/similar drugs;
2. Frequent use of sedatives, sleeping pills or other addictive drugs; History of drug abuse within 12 months prior to first administration or drug abuse screening positive;
3. Alcoholic or often drinkers within 6 months prior to screening, the average drinking amount is more than 14 units a week (1 unit= 360 ml beer or 45 ml alcohol content of 40% spirits or 150 ml wine), a heavy smoker or quitting time less than 3 months, alcohol breath test positive and nicotine test positive, and can't quit smoking and alcohol during the study;
4. Use any prescription drug or herbal tonic within one month before the first dose; Use any over-the-counter (OTC) or food supplement (including vitamins, calcium tablets, etc.) within 2 weeks before the first dose; Use of birth control pills within two weeks prior to first administration;
5. Those who have participated in other clinical trials and taken the research drugs within 3 months before the first drug administration;
6. Blood donation within 3 months before the first drug administration (including component blood donation) or blood loss greater than 400 mL, blood donation within 1 month before screening (including component blood donation) or blood loss greater than 200 mL, or receiving blood transfusion；
7. A history of autonomic dysfunction and/or a history of present illness (e.g., recurrent episodes of syncope, palpitations, etc.) within 3 years prior to first administration;
8. Previous medical history of cardiovascular, liver, kidney, lung, digestive tract, nervous system diseases, etc., which may significantly affect the absorption, distribution, metabolism and excretion of drugs, or may pose a hazard to the subjects participating in the study. The following medical history or conditions should be considered: inflammatory gastroenteritis, gastroesophageal reflux, gastrointestinal or rectal bleeding; History of pancreatic injury or pancreatitis; Greater surgical history such as gastrectomy, gastroenterostomy, or enterectomy; History of acute and chronic renal insufficiency, history of renal transplantation;
9. A history of severe vomiting and diarrhea in the previous week;
10. Female subjects during pregnancy and lactation, and female subjects of child-bearing age who cannot use contraception as required;
11. Hepatitis B surface antigen positive, hepatitis C2 antibody positive, syphilis antibody positive, HIV antibody positive;
12. Those who have special dietary requirements and cannot comply with the diet provided and the corresponding regulations;
13. Subjects refused to stop using any beverage or food containing methyl xanthine, such as coffee, tea, cola, chocolate, etc. from 48 hours before the first administration until the end of the study;
14. Subjects refused to stop using any drink or food containing grapefruit 7 days before the first dose until the end of the study;
15. Difficulty in venous blood collection or inability to tolerate venipuncture;
16. Other factors (including but not limited to inability to understand the requirements of the study, poor compliance, physical weakness, etc.) that are not suitable for participating in the study, as judged by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-05-24 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of SHR1459 | through study completion, an average of 23 days
  Peak Plasma Concentration (Cmax) of SHR1459
Pharmacokinetics parameter: AUC of SHR1459 | through study completion, an average of 23 days
  Area under the plasma concentration versus time curve (AUC) of SHR1459

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax of SHR1459 | through study completion, an average of 23 days
  Time of maximum observed concentration (Tmax) of SHR1459
Pharmacokinetics parameter: T1/2 of SHR1459 | through study completion, an average of 23 days
  Half time (T1/2) of SHR1459
Pharmacokinetics parameter: CL/F of SHR1459 | through study completion, an average of 23 days
  Total body clearance for extravascular administration (CL/F) of SHR1459
Pharmacokinetics parameter: Vz/F of SHR1459 | through study completion, an average of 23 days
  Volume of distribution (Vz/F) of SHR1459
Number of patients with Adverse Events (AEs) | through study completion, an average of 23 days
  To assess the adverse events according to CTCAE5.0
Vital sign (Blood pressure [BP]) | through study completion, an average of 23 days
  To assess the vital signs as a criteria of safety and tolerability variables.
Vital sign (pulse) | through study completion, an average of 23 days
  To assess the vital signs as a criteria of safety and tolerability variables.
Vital sign (temperature) | through study completion, an average of 23 days
  To assess the vital signs as a criteria of safety and tolerability variables.
Resting and digital electrocardiograms (ECGs) | through study completion, an average of 23 days
  To assess the cardiovascular system functioning as a criteria of safety and tolerability variables.
Physical examination | through study completion, an average of 23 days
  To assess the physical conditions as a criteria of safety and tolerability variables.
Laboratory assessments | through study completion, an average of 23 days
  To assess the hematology, clinical chemistry and urinalysis as a criteria of safety and tolerability variables.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, M.D., Ph.D., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical College, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No